CLINICAL TRIAL: NCT01002664
Title: A Phase III, Double-Blind, Randomized, Placebo-Controlled Study to Investigate the Efficacy and Safety of MCS-2 in Treating Lower Urinary Tract Symptoms Suggestive of Benign Prostatic Hyperplasia in Treatment Naïve Male Subjects
Brief Title: Efficacy and Safety of MCS-2 in the Treatment of Lower Urinary Tract Symptoms
Acronym: MCS_LUTS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Health Ever Bio-Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MCS-2-TWN-a
Record Dates: First submitted 2009-10-20; First posted 2009-10-27 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Lower Urinary Tract Symptoms; Benign Prostatic Hyperplasia
Keywords: Benign Prostatic Hyperplasia; Multi-carotenoids; MCS-2; Lower Urinary Tract Symptoms; International prostate symptom scores
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Prostatic Hyperplasia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MCS-2 (Active Comparator): Drug Name: MCS-2 Dosage: 2 soft-gel capsules Frequency: Qd per day after dinner Duration: 12 weeks
  Interventions: Drug: MCS-2
- Placebo (Placebo Comparator): Drug Name: MCS-2 placebo Dosage: 2 soft-gel capsules Frequency: Qd per day after dinner Duration: 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MCS-2 — 30 mg/day (two 15 mg capsules) Qd for 12 weeks
  Other Names: MUS
  Arms: MCS-2
Drug: Placebo — 2 soft-gel placebo capsules Qd for 12 weeks
  Other Names: MCS Matching Placebo
  Arms: Placebo

SUMMARY:
The hypothesis of the study is to examine whether MCS-2 is safe and effective in the treatment of lower urinary tract symptoms suggestive of benign prostatic hyperplasia.

DETAILED DESCRIPTION:
Eligible male subjects will be randomized to receive either MCS-2 or placebo for 12 weeks. Subjects are those not currently on any medicines for BPH or LUTS. During and at the end of the 12-week treatment period, randomized subjects will be evaluated for efficacy and safety parameters. All subjects will be advised to maintain a normal diet, similar to what was consumed before joining the study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≧ 40 years old.
* Not being treated for BPH or LUTS.
* PSA ≦ 4 ng/ml and no pathologically-proven prostate cancer.
* I-PSS ≥ 10
* No known malignancy
* AST/ALT ≦ 3X UNL.
* Creatinine ≦ 3X UNL.
* Subjects who sign the informed consent form.

Exclusion Criteria:

* Subjects' LUTS are not BPH-related
* Have been treated with pelvis irradiation or pelvic surgery.
* Plan to undergo any invasive procedures within the study period.
* Active infection or inflammation.
* Considered ineligible by the investigators.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2010-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Changes in total International Prostate Symptom Scores (I-PSS) | 12 weeks
  Changes in total International Prostate Symptom Scores (I-PSS)

SECONDARY OUTCOMES:
Changes in I-PSS subscores | 12 weeks
  Changes in I-PSS subscores
Changes in I-PSS quality of life index | 12 weels
  Changes in I-PSS quality of life index
Changes in urinary peak flow rate | 12 weeks
  Changes in urinary peak flow rate
Incidence of treatment-emergent adverse events | 12 weeks
  Incidence of treatment-emergent adverse events
Incidence of withdrawals due to treatment-emergent adverse events | 12 weeks
  Incidence of withdrawals due to treatment-emergent adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Yeong-Shiau Pu, MD PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No